CLINICAL TRIAL: NCT02968563
Title: A Prospective, Open-Label, Multicenter, Phase 2 Trial to Evaluate the Safety and Efficacy of the Combination of Tirabrutinib (GS-4059) and Idelalisib With and Without Obinutuzumab in Subjects With Chronic Lymphocytic Leukemia
Brief Title: Study to Evaluate the Safety and Efficacy of the Combination of Tirabrutinib and Idelalisib With and Without Obinutuzumab in Adults With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-401-1958; 2015-003909-42 (EudraCT Number); CLLRUmbrella1 (Other: German CLL Study Group)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tirabrutinib; idelalisib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirabrutinib + Idelalisib (Experimental): Tirabrutinib 80 mg (4 x 20 mg tablets/2 x 40 mg tablets/1 x 80 mg tablet) once daily + idelalisib 100 mg (1 x 100 mg tablet) once daily for up to 104 weeks.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Tirabrutinib + Idelalisib + Obinutuzumab (Experimental): Tirabrutinib 80 mg (4 x 20 mg tablets/ 2 x 40 mg tablets/ 1 x 80 mg tablet) once daily + idelalisib 100 mg (1 x 100 mg tablet) once daily for up to 104 weeks + obinutuzumab 100 mg on Day 1, 900 mg on Day 1 or 2, and 1000 mg subsequently for up to 8 doses on Day 1 of Weeks 2, 3, 5, and then every 4 weeks through Week 21.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Tirabrutinib — Tablets administered orally
  Other Names: GS-4059
Drug: Idelalisib — Tablets administered orally
  Other Names: Zydelig®; GS-1101; CAL-101
Drug: Obinutuzumab — Administered intravenously
  Other Names: Gazyvaro®; Gazyva®; GA101
  Arms: Tirabrutinib + Idelalisib + Obinutuzumab

SUMMARY:
The primary objective of this study is to determine the preliminary efficacy of the combination of tirabrutinib and idelalisib with obinutuzumab in adults with relapsed or refractory chronic lymphocytic leukemia (CLL).

The study has a 6 participant per arm safety run-in to evaluate safety prior to the enrollment of subsequent participants. The treatment period is adaptive, with a duration of active treatment up to two years and a total follow-up on study for up to 30 days post end of treatment, or up to Week 25 should a participant discontinue treatment prior to Week 25 for reasons other than disease progression.

ELIGIBILITY:
Key Inclusion Criteria:

* Documentation of relapsed or refractory CLL
* Requiring treatment per modified International Workshop on CLL (IWCLL) 2008 criteria; individuals without radiographically measurable disease (defined as ≥ 1 lesion > 1.5 centimetre (cm) in diameter as assessed by computed tomography (CT) or magnetic resonance imaging [MRI]) must have bone marrow evaluation at screening
* Adequate hematologic function: platelet count ≥ 50 × 10^9/L, neutrophil count ≥ 1 × 10^9/L, hemoglobin ≥ 8 grams per decilitre (g/dL) unless lower values are directly attributable to documented bone marrow burden of CLL
* Creatinine clearance (CrCl) ≥ 50 milliliter per minute (mL/min)
* Total bilirubin ≤ 1.5× institutional upper limit of normal (ULN) unless attributed to Gilbert's syndrome and aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 × ULN
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* Absence of active human immunodeficiency virus (HIV), hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, and cytomegalovirus (CMV) infection
* Satisfies the following criteria:

  * For females of childbearing potential, willingness to abstain from sexual intercourse or use a protocol-specified method of contraception as described in the study protocol
  * Males of reproductive potential who engage in sexual intercourse must agree to use protocol-specified method(s) of contraception as described in the study protocol
* Able to comply with study procedures and restrictions including mandatory prophylaxis for Pneumocystis jirovecii pneumonia (PJP)

Key Exclusion Criteria:

* Known transformation of CLL (ie, Richter's transformation, prolymphocytic leukemia)
* Known central nervous system (CNS) involvement
* Progression on treatment with any inhibitor of Bruton's tyrosine kinase (BTK), spleen tyrosine kinase (SYK), phosphatidylinositol 3-kinase (PI3K), B-cell lymphoma 2 (BCL-2), or obinutuzumab. The treatment and disease response history of individuals with prior treatment with agents in these classes should be reviewed by the sponsor or the German CLL Study Group (GCLLSG) study office prior to enrollment to clarify sensitivity to these treatments.
* Any treatment for CLL other than corticosteroids for symptomatic management within 28 days of the start of study treatment
* Participation on a concurrent therapeutic clinical trial unless all treatment is complete with only ongoing surveillance
* Diagnosis of or concern for progressive multifocal leukoencephalopathy
* History of myelodysplastic syndrome or another malignancy other than CLL, except for the following: any malignancy that has been in complete remission for 3 years, adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to start of study therapy
* Active infection requiring systemic therapy
* Pregnant or nursing women (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment and monthly during therapy)
* Active autoimmune disease or the need for higher than prednisone 10 mg daily unless for management of CLL symptoms
* Treatment or prophylaxis for CMV within the past 28 days
* History of stroke or intracranial hemorrhage within 12 months of randomization; patients requiring therapeutic anticoagulation for any indication should be discussed with the GCLLSG cooperating physician and/or medical monitor prior to screening.
* Use of a strong CYP3A4 or a strong P-glycoprotein (P-gp) inducer within 2 weeks of first dose of study treatment or anticipated chronic use while on study
* Demonstration of corrected QT (QTc) interval > 450 milliseconds or requirement for ongoing treatment with concomitant medications that prolong the QT interval

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (14):
- Germany (14):
  - Ambulante Krebszentrum Schaubstraße, Frankfurt (Oder), Brandenburg
  - Hämatologische-onkologische Gem.-Praxis Dres. Brudler-Heinrich-Bangerter, Augsburg, Augsburg
  - Uniklinik Koln, Cologne
  - Internistische Gemeinschaftspraxis Dres. Schliesser-Käbisch-Weber, Gießen, Giessen
  - Uniklinik Leipzig, Leipzig
  - Luebecker Onkologische Schwerpunktpraxis, Lübeck
  - Universitasmtedizin Mannheim, Mannheim
  - KH Maria Hilf-Franziskushaus, Mönchengladbach, Mönchengladbach
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Krankenhaus München-Schwabing, München
  - Klinikum Rechts der Isar der Technischen Universität München, München
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Facharztzentrum Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany. The first participant was screened on 13 December 2016. The last study visit occurred on 14 January 2021.
Pre-assignment Details: 35 participants were screened. Randomization was discontinued after implementation of Protocol Amendment 3; all additional participants were enrolled to Arm: Tirabrutinib + Idelalisib + Obinutuzumab.
Groups:
- Tirabrutinib + Idelalisib: Tirabrutinib 80 mg (4 x 20 mg tablets/2 x 40 mg tablets/1 x 80 mg tablet) orally once daily + idelalisib 100 mg (1 x 100 mg tablet) orally once daily for up to 104 weeks.
- Tirabrutinib + Idelalisib + Obinutuzumab: Tirabrutinib 80 mg (4 x 20 mg tablets/ 2 x 40 mg tablets/ 1 x 80 mg tablet) orally once daily + idelalisib 100 mg (1 x 100 mg tablet) orally once daily for up to 104 weeks + obinutuzumab 100 mg on Day 1, 900 mg on Day 1 or 2, and 1000 mg subsequently for up to 8 doses on Day 1 of Weeks 2, 3, 5, and then every 4 weeks through Week 21.
Period: Overall Study
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Started | 5 | 30
Completed | 4 | 22
Not Completed | 1 | 8
Not completed — Adverse Event | 0 | 6
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized or enrolled participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab | Total
Number analyzed (Participants) | 5 | 30 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (4.7) | 65 (9.4) | 65 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 2 | 20 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: White | 5 | 29 | 34
    Race: Not Permitted | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 5 | 29 | 34
    Ethnicity: Not Permitted | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response/Complete Remission (CR), as Assessed by Investigator Using Modified International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Criteria at Week 25
Description: Rate of CR per modified IWCLL 2008 criteria at Week 25 was defined as the percentage of participants who achieved CR/complete remission with incomplete recovery of the bone marrow (CRi) at Week 25. CR: meeting following criteria and no disease related symptoms: no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow sample must be normocellular with 30% lymphocytes and no B-lymphoid nodules; platelets > 100,000/µL; hemoglobin > 11 g/dL; and neutrophils > 1500/µL. CRi: CR criteria (no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow [hypocellular] with 30% lymphocytes and no B-lymphoid nodules), persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity.
Time Frame: Week 25
Population: The Full Analysis Set included all randomized or enrolled participants who received at least 1 dose of any study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Number analyzed (Participants) | 5 | 30
percentage of participants | 0 [0 to 45.1] | 6.7 [1.2 to 19.5]

2. Secondary Outcome: Rate of CR With Bone Marrow Minimal Residual Disease (CR/BM MRD) Negativity, as Assessed by the Investigator Using the Modified IWCLL 2008 Criteria at Week 25
Description: Rate of CR/BM MRD at Week 25 was defined as percentage of participants who achieved CR/CRi per modified IWCLL 2008 criteria and also achieved BM MRD negativity at Week 25. CR: meeting following criteria and no disease related symptoms: no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow sample must be normocellular with 30% lymphocytes and no B-lymphoid nodules; platelets > 100,000/µL; hemoglobin > 11 g/dL; and neutrophils > 1500/µL. CRi: CR criteria (no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow [hypocellular] with 30% lymphocytes and no B-lymphoid nodules), persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. MRD response was assessed with four-color-flow cytometry (FACS) and MRD negativity was defined as one CLL cell per 10,000 leukocytes [0.01%], ie,<10^-4 and participants were defined as MRD negative if their disease burden was below this threshold.
Time Frame: Week 25
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Number analyzed (Participants) | 5 | 30
percentage of participants | 0 [0 to 45.1] | 0 [0 to 9.5]

3. Secondary Outcome: Rate of CR With Peripheral Minimal Residual Disease (CR/PB MRD) Negativity, as Assessed by the Investigator Using the Modified IWCLL 2008 Criteria at Week 25
Description: Rate of CR/PB MRD at Week 25 was defined as the percentage of participants who achieved CR/CRi per modified IWCLL 2008 criteria and also achieved PB MRD negativity at Week 25. CR: meeting following criteria and no disease related symptoms: no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow sample must be normocellular with 30% lymphocytes and no B-lymphoid nodules; platelets > 100,000/µL; hemoglobin > 11 g/dL; and neutrophils > 1500/µL. CRi: CR criteria (no lymphadenopathy > 1.5 cm/hepatomegaly/splenomegaly; lymphocytes < 4000/μL; bone marrow [hypocellular] with 30% lymphocytes and no B-lymphoid nodules), persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. MRD response was assessed with FACS and MRD negativity was defined as one CLL cell per 10,000 leukocytes [0.01%], ie,<10^-4 and participants were defined as MRD negative if their disease burden was below this threshold.
Time Frame: Week 25
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Number analyzed (Participants) | 5 | 30
percentage of participants | 0 [0 to 45.1] | 0 [0 to 9.5]

4. Secondary Outcome: Overall Response Rate (ORR), as Assessed by the Investigator Using the Modified IWCLL 2008 Criteria at Week 25
Description: ORR was assessed based on modified IWCLL 2008 criteria and was defined as percentage of participants achieving a CR, CRi, partial remission (PR; including nodular partial response [nPR]), and PR with lymphocytosis (PR-L). CR and CRi: meeting all the criteria that have been defined in Outcome measures 1, 2 and 3. PR: ≥ 2 of these: ≥ 50% decrease in lymphocytes, lymphadenopathy, size of liver, size of spleen, and 50% decrease in bone marrow infiltrates; and ≥ 1 of these: neutrophils > 1500/μL or ≥ 50% increase from Baseline, platelets ≥ 100,000/µL or ≥ 50% increase from Baseline, hemoglobin >11 g/dL or ≥ 50% increase from Baseline. PR-L: meeting PR criteria; however, a lymphocytosis related to treatment may be present. nPR: All criteria for a CR/CRi were fulfilled, but the bone marrow showed lymphoid nodules.
Time Frame: Week 25
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Number analyzed (Participants) | 5 | 30
percentage of participants | 60.0 [18.9 to 92.4] | 93.3 [80.5 to 98.8]

5. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: Treatment-emergent AEs are defined as 1 or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
  * Any AEs leading to discontinuation of study drug
  A SAE is defined as an event that, at any dose, resulted in any of the following: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or a medically important event or reaction.
Time Frame: First dose date up to the last dose date (maximum: 105 weeks) plus 30 days
Population: The Safety Analysis Set included all randomized or enrolled participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
Number analyzed (Participants) | 5 | 30
percentage of participants
  Any Treatment-Emergent AEs | 100 | 100
  Treatment-Emergent SAEs | 60.0 | 46.7

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (maximum: 105 weeks) plus 30 days; All-Cause Mortality: Enrollment up to 31 months
Description: Adverse Events: The Safety Analysis Set included all randomized or enrolled participants who received at least 1 dose of any study drug.
  All-Cause Mortality: The All Enrolled Analysis Set included all participants who received a study participant identification number in the study after screening.
Groups:
- Tirabrutinib + Idelalisib + Obinutuzumab: Tirabrutinib 80 mg (4 x 20 mg tablets/ 2 x 40 mg tablets/ 1 x 80 mg tablet) orally once daily + idelalisib 100 mg (1 x 100 mg tablet) orally once daily for up to 104 weeks + obinutuzumab 100 mg on Day 1, 900 mg on Day 1 or 2, and 1000 mg subsequently for up to 8 doses administered intravenously over 21 weeks.
Arm/Group | Tirabrutinib + Idelalisib | Tirabrutinib + Idelalisib + Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/30
Serious Adverse Events (participants affected / at risk) | 3/5 | 14/30
Other Adverse Events (participants affected / at risk) | 5/5 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirabrutinib + Idelalisib (N=5) | Tirabrutinib + Idelalisib + Obinutuzumab (N=30)
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Large intestine infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tirabrutinib + Idelalisib (N=5) | Tirabrutinib + Idelalisib + Obinutuzumab (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8
Tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 6
Lacrimation increased (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 2
Visual impairment (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 10
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 7
Vomiting (Gastrointestinal disorders) | 1 | 4
Chills (General disorders) | 1 | 6
Fatigue (General disorders) | 1 | 10
Feeling cold (General disorders) | 0 | 2
Influenza like illness (General disorders) | 0 | 2
Medical device pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 7
Bronchitis (Infections and infestations) | 0 | 6
Conjunctivitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 0 | 2
Herpes virus infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 10
Oral pustule (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 7
Urinary tract infection (Infections and infestations) | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 5
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
C-reactive protein increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 0 | 3
Weight decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 4
Memory impairment (Nervous system disorders) | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3
Haematoma (Vascular disorders) | 1 | 6
Hypertension (Vascular disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02968563/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02968563/SAP_003.pdf